CLINICAL TRIAL: NCT06710587
Title: A Decentralised Open Label Trial to eValuate the Efficacy Of the VoY Program in A Patient Population Using GLP/GIP-1RA thERapy
Brief Title: Does Use of the Voy Program Improve Weight Loss Percentage and Other Health Outcomes in a Population Already Taking GLP/GIP-1RA Medication?
Acronym: VOYAGER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Menwell Limited (Industry)
Collaborators: Lindus Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LH-MAN-01; 350648 (Other: IRAS)
Record Dates: First submitted 2024-11-22; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Obesity; Weight Loss
Keywords: Voy Program
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Open label, parallel-group, superiority randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - Standard Pathway (No Intervention): Standard GLP/GIP-1RA pathway as offered by Voy as part of participants usual care for weight loss
- Intervention - Standard Pathway + Voy Program (Experimental): Standard GLP/GIP-1RA pathway as offered by Voy as part of participants usual care for weight loss + Voy Program - coaching and access to the Voy app to support behavioural changes
  Interventions: Behavioral: Voy Program

INTERVENTIONS:
Behavioral: Voy Program — Voy Program - coaching and access to the Voy app to support behavioural changes
  Arms: Intervention - Standard Pathway + Voy Program

SUMMARY:
The aim of the trial is to assess the impact of the Voy Program on weight loss and other health outcomes in an obese population already approved for GLP/GIP-1RA medication.

If an eligible participant consents to take part in the trial, they will be randomly allocated into one of the two trial groups. One group will continue with the standard pathway for GLP/GIP-1RA as part of their usual care for weight loss, while the other group will utilise the Voy Program in addition to the standard pathway.

In the intervention group, the Voy Program will include personalised sessions with a qualified coach as well as access to resources including managing nutrition and movement. The frequency of the coaching sessions will be led by the participant but will normally start fortnightly.

All participants will be enrolled in the trial for 12 months and will be asked to complete questionnaires on a monthly and quarterly basis.

DETAILED DESCRIPTION:
This is a decentralised, single site, open label, parallel-group, superiority randomised controlled trial in participants with a BMI ≥30 (or BMI ≥27 with certain comorbidities) already offered GLP/GIP-1RA through Voy's standard pathway as part of their usual care for weight loss. A total of 470 eligible participants will be randomised in the UK to receive the standard pathway (GLP/GIP-1RA only - control arm), or the standard pathway (GLP/GIP-1RA) plus the Voy Program (intervention arm).

Screening, informed consent and eligibility assessments will occur online. Participants in the intervention group will receive coaching sessions via video and phone calls with a qualified coach. These sessions will be participant led but will normally initially occur fortnightly. Participants in the intervention arm will also have access to all available features in the Voy app, which is used to book coaching sessions and also includes content around nutrition and exercise management, weight progress tracking, and an AI-powered meal analysis tool to support behavioural changes. Participants will be expected to complete surveys monthly. Participants will enter data directly into the trial web platform, EDC platform or the sponsors platform (Voy). Participation in the initial trial is expected to last approximately 12 months, with optional long term follow-up continuing for an additional 12 months (24 months total).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65.
2. BMI≥30,

   a. Or BMI≥27 with any of the following comorbidities as diagnosed by a Doctor:
   * High blood pressure
   * High cholesterol
   * Obstructive sleep apnoea
   * Erectile dysfunction
   * Asthma
   * Osteoarthritis
   * Chronic back pain
   * PCOS
   * Fatty liver disease
3. Approved for the standard GLP/GIP-1RA pathway by Voy as part of usual care for weight loss.
4. People who use either an iOS or Android smartphone using operating system iOS 16 or Android 8 or later.
5. Agree to not use another intervention for weight loss for the duration of the trial.

   * Other diet specific interventions such as meal replacement shakes.
   * Over the counter medication / supplements such as appetite suppressants, thermogenics, herbal supplements.
   * Any other medicated weight loss program.
   * Structured weight loss programs such as Weight Watchers, Noom, Second Nature.
   * Non-surgical medical weight management such as lipotropic injections and metabolic enhancers.
   * Surgical interventions such as a gastric bypass, banding, or other bariatric surgery
   * Other personalised nutrition programmes, such as ZOE
6. Able and willing to provide Informed Consent and adhere to trial procedures.

Exclusion Criteria:

1. Pregnant or breastfeeding women, or those planning to get pregnant in the next 12 months.
2. Known diabetes mellitus (Type 1 or 2) or thyroid disease.
3. Previous surgery or endoscopic intervention for obesity, or planned surgery or endoscopic intervention for obesity in the next 12 months.
4. Lost ≥ 5kg in the last 3 months intentionally or otherwise.
5. Currently using other weight loss medications, or use of other weight loss medications in the past 6 months.
6. Currently using medications that cause weight gain, including systemic steroids, or used such medications in the past 6 months.
7. Severe anxiety or depression (either PHQ-9 >15 or GAD7 >10).
8. Severe eating disorder (Binge eating scale ≥27).
9. Participation in another interventional clinical study or use of investigational drugs in the last 6 months.
10. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2025-01-02 (Estimated); Primary Completion 2026-04-02 (Estimated); Study Completion 2027-04-02 (Estimated)

PRIMARY OUTCOMES:
Percentage weight loss Percentage weight loss | Primary endpoint of 12 months; with data collected at Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  To evaluate and draw inferences on the percentage weight loss in participants prescribed GLP/GIP-1RA therapy with and without the Manual Voy Program

SECONDARY OUTCOMES:
Absolute and percentage change in waist to height ratio | Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  To evaluate the impact of the Voy Program on waist to height ratio over 12 months
Absolute and percentage change in waist to hip ratio | Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  To evaluate the impact of the Voy Program on waist to hip ratio over 12 months
Absolute and percentage change in Blood glucose (HbA1c) and CRP | Baseline, Months 3, 6, 9, 12
  To evaluate the impact of the Voy Program on Metabolic parameters over 12 months
Absolute and percentage change in Lipid profile (total cholesterol, LDL, HDL, triglycerides) | Baseline, Months 3, 6, 9, 12
  To evaluate the impact of the Voy Program on Metabolic parameters over 12 months
Absolute and percentage change in CRP | Baseline, Months 3, 6, 9, 12
  To evaluate the impact of the Voy Program on Metabolic parameters over 12 months
Change in blood pressure | Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  To evaluate the impact of the Voy Program on Vital signs over 12 months
Change in heart rate | Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  To evaluate the impact of the Voy Program on Vital signs over 12 months
Change in Comorbidity status (i.e. new diagnosis) | Baseline, Months 3, 6, 9, 12
  To evaluate the impact of the Voy Program on the status of obesity-related comorbidities at 12 months, such as hypertension, dyslipidemia and progression to raised / abnormal HbA1C
Change in patient activation measured using the following validated questionnaire: Patient Activation Measure-10 (PAM-10) | Baseline, Months 3, 6 9, 12
  To evaluate the impact of the Voy Program on Patient Activation 12 months - a higher score = a higher activation level (0-100)
Change in quality of life measured using the following validated questionnaires: EQ-5D-5L | Baseline, Months 3, 6 9, 12
  To evaluate the impact of the Voy Program on Quality of life at 12 months (level 1-5 with 1 being no problems and 5 being extreme problems)
Change in health and quality of life measured using the following unvalidated questionnaires: Voy's weight-related quality of life survey | Baseline, Months 3, 6 9, 12
  To evaluate the impact of the Voy Program on Quality of life at 12 months - questions use 5-part likert scale with 1 being no problems/never, and 5 being lots of problems/always
Changes in Body fat percentage measured via Renpho bluetooth scale | Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  To evaluate the impact of the Voy Program on Body fat percentage over 12 months
Changes in anxiety using scores derived from validated questionnaire Generalised Anxiety Disorder-7 item (GAD-7) | Baseline, Months 3, 6 9, 12
  To evaluate the impact of the Voy Program on anxiety over 12 months (The cut-off points for mild, moderate, and severe anxiety are 5, 10, and 15, respectively)
Changes in mental health using scores derived from validated questionnaire The Patient Health Questionnaire (PHQ-9) | Baseline, Months 3, 6 9, 12
  To evaluate the impact of the Voy Program on mental health over 12 months (The PHQ-9 score ranges from 0 to 27, with the following ranges indicating the severity of depression:
  0-4: None or minimal depression 5-9: Mild depression 10-14: Moderate depression 15-19: Moderately severe depression 20-27: Severe depression)
Changes in eating disorders using scores derived from validated questionnaire Binge Eating Scale (BES) | Baseline, Months 3, 6 9, 12
  To evaluate the impact of the Voy Program on eating disorders over 12 months (no binge eating (score ≤ 17), mild to moderate binge eating (score of 18 - 26) and severe binge eating (score ≥ 27))
Changes in eating disorders using scores derived from validated questionnaire The Three Factor Eating Questionnaire (TFEQ-R18) | Baseline, Months 3, 6 9, 12
  To evaluate the impact of the Voy Program on eating disorders over 12 months (Higher scores indicate more Uncontrolled, Restraint and Emotional eating)
Occurrence of (serious) adverse events. | Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  To evaluate the impact of the Voy Program on occurrence of (S)AEs throughout the trial
Cost-utility analysis on healthcare utilisation questionnaire | Baseline, Months 3, 6 9, 12
  To evaluate the impact of the Voy Program on Health Economic Outcomes and productivity over 12 months
Maintenance of weight loss at 24 months | Month 24
  To evaluate the impact of the Voy Program on long-term outcomes (weight loss maintenance) over 24 months
Changes in diet quality | Baseline, Months 3, 6 9, 12
  Changes in diet quality using scores derived from the following validated questionnaire: Rapid Prime Diet Quality Score Screener (rPDQS) - (scoring is a traffic light logic system (green= healthy dietary pattern; yellow = less healthy dietary pattern; red = unhealthy dietary pattern), assigning 0 points for red, 1 for yellow, and 2 for green-coded frequency of food group consumption, with a potential range of 0 to 26)

CONTACTS AND LOCATIONS:
Overall Officials: Carel Le Roux, Principal Investigator — Ulster University; Werd Al-Najim, Principal Investigator — Ulster University

IPD SHARING:
Plan to Share IPD: No